CLINICAL TRIAL: NCT04912453
Title: A Randomised Controlled Trial to Compare Primary Anastomosis Versus Enterostomy in the Surgical Treatment of Necrotising Enterocolitis
Brief Title: Primary Anastomosis Versus Enterostomy in the Surgical Treatment of Necrotising Enterocolitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NECHKTrial
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-05

CONDITIONS: Necrotizing Enterocolitis
Keywords: Necrotizing Enterocolitis; Neonatal surgery; Primary anastomosis; Enterostomy
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Enterostomy

STUDY DESIGN:
Intervention Model Description: All neonates with confirmed NEC and require surgical intervention will be included. This is a local multi-centre study and neonates from the three centres which perform neonatal surgery will participate. At laparotomy, the diseased segment of intestine will be resected and the patients will then receive either primary anastomosis or enterostomy according to randomisation done pre-operatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary anastomosis group (Experimental)
  Interventions: Procedure: Primary anastomosis
- Enterostomy group (Experimental)
  Interventions: Procedure: Enterostomy

INTERVENTIONS:
Procedure: Primary anastomosis — At laparotomy, the diseased segment of intestine will be resected and the patients will then receive primary anastomosis
  Arms: Primary anastomosis group
Procedure: Enterostomy — At laparotomy, the diseased segment of intestine will be resected and the patients will then receive enterostomy
  Arms: Enterostomy group

SUMMARY:
Necrotizing enterocolitis (NEC) is a devastating disease that affects the intestine of premature infants and is the most common surgical emergency in newborns. It is estimated that up to 10% of premature babies can suffer from this condition. Despite aggressive medical treatment, surgical intervention is necessary in up half of the cases for bowel necrosis or perforation and these often represent the more severe form of the disease. The advances in neonatal intensive care and surgical knowledge have resulted in improved survival rate in recent years.

For NEC patients with severe disease (i.e.) those with intestinal perforation or gangrenous bowel not responding to medical therapy, surgery with resection of diseased segments is the treatment of choice. Traditional surgical approach would be to resect the diseased bowel segment with formation of enterostomy. However, in a few advanced centres, primary anastomosis after the resection of diseased bowel segment is practised. Retrospective reports of the primary anastomosis approach have shown that this is also a viable option with no increased rate of peri-operative morbidity. It also has the advantage of avoiding a second operation for enterostomy closure. Nonetheless, prospective studies comparing the two approaches are lacking.

The proposed study will fill up the following knowledge gap on what the best surgical option for NEC at laparotomy is. The findings will help guide our practice for NEC patients in the future in order to provide them with the best possible and evidence-based care.

In this study, the investigators hypothesize that neonates with major NEC undergoing primary anastomosis after surgical resection is not inferior to neonates who have enterostomy, in terms of peri-operative morbidities.

Aim of the study is to compare the short term and medium term outcomes of NEC patients requiring surgical intervention who either receive primary anastomosis or enterostomy creation.

ELIGIBILITY:
Inclusion Criteria:

* All neonates with confirmed NEC and require surgical intervention will be included

Exclusion Criteria:

1. Neonates found to have NEC totalis and deemed unsalvageable;
2. Neonates found to have multiple sites of gangrenous bowels which require more than two anastomoses;
3. Neonates found to be extremely unstable cardiovascularly intra-operatively and can only withstand excision of gangrenous bowels, but will not allow anastomosis or stoma creation;
4. Parents who do not agree to participate in the study
5. Neonates found to have pathology other than NEC after recruitment (either on intraoperative findings or pathological findings on surgical specimens).

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Re-operation rate of the two surgical approaches | 6 months

SECONDARY OUTCOMES:
Wound-related problems | 6 months
  Wound problems not requiring re-operations e.g. wound infection; stomal prolapse; incisional hernia
Time to full enteral feeding | 6 months
  Time needed (in term of days) to achieve full enteral feeding (defined as 150ml/kg/day) and stoppage of parenteral feeding

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth KY Wong, MD, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Surgery, University of Hong Kong, Hong Kong, Hong Kong